CLINICAL TRIAL: NCT03488290
Title: Building Resilience Against ViolencE (BRAVE): A Parenting Intervention for Mothers and Fathers With Post-traumatic Stress Symptoms.
Brief Title: Building Resilience Against ViolencE (BRAVE)
Acronym: BRAVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PILL-BRAVE01
Record Dates: First submitted 2018-03-28; First posted 2018-04-04 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Parents; Young Children; Trauma Focused Cognitive Behavior Therapy; Learning Through Play
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Long-Term Potentiation; Therapeutics

STUDY DESIGN:
Intervention Model Description: This will be a two arm study: 1) LTP Plus TF-CBT added to TAU 2) Treatment as usual (TAU)
Who Masked: Outcomes Assessor
Masking Description: Researchers doing outcome assessment will be kept blind to the group allocations
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LTP Plus TF CBT (Experimental): LTP Plus TF CBT group participants will receive group intervention by masters' level trained facilitators weekly during the first two months and then fortnightly. It comprises of two components i.e. LTP and TF CBT. LTP aims at enabling parents to improve their child's psychosocial development by educating about child development and the importance of mother-child play. TF CBT aim is to modify excessively negative appraisals of the trauma and its sequelae by careful questioning
  Interventions: Behavioral: LTP Plus TF-CBT; Other: Treatment as Usual
- Treatment as Usual (Other): TAU group will receive routine care consisting of routine follow ups
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: LTP Plus TF-CBT — Experimental: LTP Plus TF-CBT LTP Plus TF-CBT group participants will receive group intervention by masters' level trained facilitators weekly during the first two months and then fortnightly. It comprises of two components i.e. LTP and TF CBT. LTP aims at enabling parents to improve their child's psychosocial development by educating about child development and the importance of mother-child play. TF CBT aim is to modify excessively negative appraisals of the trauma and its sequelae by careful questioning
  Arms: LTP Plus TF CBT
Other: Treatment as Usual — The Treatment as Usual group will receive routine care

SUMMARY:
The study has both quantitative and qualitative components.

The objective of the quantitative study is:

To evaluate the effectiveness of Learning Through Play (LTP) Plus culturally adapted Trauma Focused Cognitive Behavior Therapy (TF-CBT) for post-traumatic stress symptoms in parents.

The objective of the qualitative study is:

To find out facilitators and barriers from the perspective of the participants and other stakeholders (e.g., clinicians, GPs, people delivering the LTP plus TF CBT intervention etc)

DETAILED DESCRIPTION:
Despite the high prevalence of post-traumatic stress disorder in Pakistan, research on psychosocial intervention is limited. We propose to investigate the acceptability, feasibility and effectiveness of manual assisted Learning Through Play (LTP) Plus culturally adapted Trauma Focused Cognitive Behavior Therapy (TF-CBT) among parents experiencing Post Traumatic Stress Disorder (PTSD). LTP Plus is proposed as a low cost intervention to improve parents' mental and physical health, and promote healthy child development. The LTP research-based activities enhance children's development while simultaneously promoting attachment security through building parents' ability to read and be sensitive to their children's cues and through active involvement in their children's development. This will be integrated with Trauma Focused CBT.

Purpose of this RCT is to determine the effectiveness of LTP plus TF- CBT intervention. The study will be conducted in two cities of Pakistan, Karachi and Peshawar.Participants will be screened using Impact of Event Scale-Revised (IES-R) and eligibility checklist. Those scoring 24 or above will be eligible for more in depth assessment. Assessments will be done at baseline and after completion of intervention. Outcome assessments will be done by independent Research Assistants blind to group allocations.

ELIGIBILITY:
Inclusion Criteria:

Participants will be included in the study if they are:

Parents over the age of 16 years who are living with their children age 3-6 years. They meet the criteria for Post-Traumatic Stress Disorder (PTSD) and are able to give informed consent

Exclusion Criteria:

Participants will be excluded from the study if they have:

Any diagnosed physical or learning disability which prevents them from attending the LTP+ group intervention, or suffering from psychosis or those who are actively suicidal. This will be assessed by the research team at screening stage. Any disabilities or diagnosed mental illness. Any parent who is on current use of anti-depressant medication. And a prior self-reported mental illness, including depression.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Clinically administered PTSD Scale-5 (CAPS-5) | Changes from Baseline to 4th Month
  The Clinical Administered PTSD Scale-5 (CAPS-5) is a 30 item scale and will be used as a primary outcome measure as this is the goal standard and structured interview for assessing post-traumatic stress disorder (PTSD), diagnostic status and symptom severity (Weathers et al., 2013).Higher score indicate greater severity.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | Changes from Baseline to 4th Month
  PHQ-9 is 10 items self-report questionnaire which is easy to use and can be administered by a trained research worker. A score of 10 or above is taken as cut -off point for depressive disorder. This scale will be used to check severity of depression.Higher score indicate greater severity of depression.
Generalized Anxiety Disorder (GAD) 7 | Changes from Baseline to 4th Month
  The GAD-7 is a seven item scale will be used to screen for and measure severity of Generalized Anxiety Disorder. Higher score indicate greater severity of anxiety.
Client Service Receipt Inventory (CSRI) | Changes from Baseline to 4th Month
  This will be used to collect information about the use of other health services (including the informal sector faith healers/Imams).
Ages and Stages Questionnaire | Changes from Baseline to 4th Month
  To assess physical, social, emotional and cognitive development of children.

CONTACTS AND LOCATIONS:
Overall Officials: Nasim Chaudhry, Principal Investigator — Pakistan Institute of Living & Learning
Locations (2):
- Pakistan (2):
  - Schools, Community, Peshawar, Khyber Pakhtunkhwa
  - Schools, Community, Karachi, Sindh

REFERENCES:
- [Background] Allen B, Lauterbach D. Personality characteristics of adult survivors of childhood trauma. J Trauma Stress. 2007 Aug;20(4):587-95. doi: 10.1002/jts.20195. PMID 17721954
- [Background] Byrne CA, Riggs DS. The cycle of trauma; relationship aggression in male Vietnam veterans with symptoms of posttraumatic stress disorder. Violence Vict. 1996 Fall;11(3):213-25. PMID 9125790
- [Background] Cartwright K, El-Khani A, Subryan A, Calam R. Establishing the feasibility of assessing the mental health of children displaced by the Syrian conflict. Glob Ment Health (Camb). 2015 Jun 19;2:e8. doi: 10.1017/gmh.2015.3. eCollection 2015. PMID 28596856
- [Background] Dubrow NF, Garbarino J. Living in the war zone: mothers and young children in a public housing development. Child Welfare. 1989 Jan-Feb;68(1):3-20. PMID 2914517
- [Background] El-Khani A, Cartwright K, Redmond A, Calam R. Daily bread: a novel vehicle for dissemination and evaluation of psychological first aid for families exposed to armed conflict in Syria. Glob Ment Health (Camb). 2016 Apr 22;3:e15. doi: 10.1017/gmh.2016.9. eCollection 2016. PMID 28596884
- [Background] El-Khani A, Ulph F, Redmond AD, Calam R. Ethical issues in research into conflict and displacement. Lancet. 2013 Aug 31;382(9894):764-5. doi: 10.1016/S0140-6736(13)61824-3. No abstract available. PMID 23993182